CLINICAL TRIAL: NCT06717217
Title: Determinating the Effect of Nursing Education Given Before Tympanoplasty Surgery on Postoperative Pain and Complications
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Muğla Sıtkı Koçman University (Other)
Responsible Party: Principal Investigator, Şeyda KORKMAZ, Master's Degree Student, Muğla Sıtkı Koçman University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MSKU-ENT-KORKMAZ-001
Record Dates: First submitted 2024-12-01; First posted 2024-12-04 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-03

CONDITIONS: Nursing Education; Postoperative Pain; Postoperative Complications; Tympanoplasty Surgery; ENT Surgery
MeSH Terms: conditions — Pain, Postoperative; Postoperative Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CONTROL GROUP (No Intervention)
- WORKING GROUP (Experimental)
  Interventions: Procedure: NURSING EDUCATION GIVEN BEFORE TYMPANOPLASTY SURGERY

INTERVENTIONS:
Procedure: NURSING EDUCATION GIVEN BEFORE TYMPANOPLASTY SURGERY — EAR CARE TRAINING
  Arms: WORKING GROUP

SUMMARY:
Health and illness are complex, universal ideas addressed from a holistic approach. Advancements in healthcare have led to an increase in life expectancy, a rise in the prevalence of chronic diseases, and an escalation in the number of surgical procedures conducted . Surgical techniques influence individuals' health and illness progression. Patients having surgical operations require the attention of nurses and other healthcare workers to address the ramifications of the procedure .

Nurses have performed numerous responsibilities in patient care. These tasks pertain to expediting recovery post-illness and maintaining health continuity. Discharge training is also incorporated into the processes implemented to meet these responsibilities. Discharge training seeks to expedite recovery and mitigate the onset of problems. Discharge training is essential for equipping surgical patients with the requisite information and abilities for post-discharge care.

Ear, Nose, and Throat (ENT) surgeries significantly influence persons' quality of life, as they impact hearing and balance, distinguishing them from other surgical interventions. Consequently, patient care and discharge education following ear surgery play a crucial role in recovery and health enhancement.

The ears serve as the organs of auditory perception and equilibrium. Tympanoplasty is performed on individuals with tympanic membrane perforations or ossicular chain injury that impairs hearing and balance. Tympanoplasty is a surgical intervention that entails the restoration of the ossicular chain (malleus, incus, stapes) and/or the installation of a fascia graft to restore auditory function.

This study aims to assess the impact of preoperative nurse education on postoperative pain and complication rates following tympanoplasty.

DETAILED DESCRIPTION:
This research will take place at the Otorhinolaryngology department of Hacettepe University Adult Hospital. The objective is to track pain progression and problems during the postoperative period through ear care instruction provided to patients prior to tympanoplasty surgery, leading to the establishment of a quasi-experimental research design. The study seeks to assess pain and complications during the early surgical phase (first 24 hours) and at the first post-discharge follow-up (subsequent interval).

Based on the calculations conducted with the G Power 3.1 program, it was determined to include 56 patients in the trial, with 28 assigned to the experimental group and 28 to the control group. The experimental group is scheduled to receive ear care instruction alongside standard preoperative treatment. The control group will receive only standard treatment without any further interventions. The postoperative period will involve an assessment of pain and complication development in both groups during the early (first 24 hours) and late (first follow-up after discharge) phases.

The postoperative pain levels of the patients will be assessed using the Visual Analog Scale (VAS). The assessment will include pain within the first 24 hours postoperatively and early complications such as hemorrhage, hematoma, hypothermia, hyperthermia, tachycardia, nausea, vomiting, hypotension, hypertension, and alveolar collapse. Subsequent complications, including pain, delayed wound healing, wound infection characterized by erythema, localized hyperthermia, edema, wound dehiscence, abscess formation, necrosis at the wound site due to insufficient nutrition and improper closure, and cellulitis, will be assessed during the initial post-discharge evaluations.

Study Hypotheses H01: Nursing education provided before to tympanoplasty surgery does not influence postoperative pain levels.

H11:Nursing education administered before to tympanoplasty surgery influences postoperative pain levels.

H02:Nursing education provided before to tympanoplasty surgery does not influence postoperative complications.

H03:Nursing education provided prior to tympanoplasty surgery influences the occurrence of postoperative problems.

ELIGIBILITY:
Criteria for Inclusion

* Patients who consented to participate in the study
* Patients with literacy skills
* Individuals aged 18 to 65 years
* Individuals who have received tympanoplasty surgery
* Patients were monitored preoperatively and postoperatively at Hacettepe University Adult Hospital.

Criteria for Exclusion:

* Patients who declined to participate in the study
* Patients receiving tympanoplasty for cholesteatoma. Assessing the progression of issues in individuals diagnosed with cholesteatoma (abnormal skin epithelial growth in the middle ear cavity) is inappropriate due to the presence of repeated perforations and aberrant tissue proliferation.
* Individuals with psychological disorders
* Patients who are foreign nationals.
* Individuals with speech impairments and irreversible hearing loss

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2024-12-05 (Estimated); Primary Completion 2024-12-25 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Development of complications | Postopreative 0.day-6.day
  These issues typically arise within the initial 24 hours post-surgery. These encompass hemorrhage/hematoma, hypothermia/hyperthermia, arrhythmia, nausea/emesis, hypotension/hypertension, and pulmonary collapse/atelectasis.
  Late complications refer to those that may arise after the third postoperative day. The complications encompass delayed wound healing, wound infection (characterized by localized temperature elevation, edema, and erythema), wound dehiscence, wound abscess, cellulitis, and psychological issues (Manekk et al., 2022).

SECONDARY OUTCOMES:
Visual Analog Scale | Postopreative 0.day-6.day
  The Visual Analog Scale (VAS) is a self-administered instrument including a horizontal or vertical line, typically 10 cm in length (100 mm), with two spoken descriptors indicating pain levels at either end. A modification in the visual analog scale score signifies a relative alteration in the intensity of the pain feeling. The patient is requested to denote their perceived pain intensity on a 100 mm horizontal line, with the measurement taken from the left edge to determine the VAS score. The VAS score exhibits a strong correlation with acute pain levels (Chiarotto et al., 2019).
  The patient is requested to evaluate their pain using a scale from 0 to 10, where 0 signifies no pain and 10 represents the most severe pain conceivable (Shafshak & Elnemr, 2021).

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ahmed Mohamed Eldesoky, H., & Mahmoud Mahmoud, H. (2019). Effect of Implementing a Nursing Management Protocol on Postoperative Health Outcomes for Patients undergoing Tympanoplasty. Egyptian Journal of Health Care, 10(4), 471-491
- [Background] Millward, K. (2017). Ear care: an update for nurses (part 2). Practice Nursing, 28(8), 332-337
- [Background] Kang E, Gillespie BM, Tobiano G, Chaboyer W. General surgical patients' experience of hospital discharge education: A qualitative study. J Clin Nurs. 2020 Jan;29(1-2):e1-e10. doi: 10.1111/jocn.15057. Epub 2019 Oct 17. PMID 31509311
- [Background] Jerofke T, Weiss M, Yakusheva O. Patient perceptions of patient-empowering nurse behaviours, patient activation and functional health status in postsurgical patients with life-threatening long-term illnesses. J Adv Nurs. 2014 Jun;70(6):1310-22. doi: 10.1111/jan.12286. PMID 24847530
- [Background] Miller MJ, Abrams MA, Earles B, Phillips K, McCleeary EM. Improving patient-provider communication for patients having surgery: patient perceptions of a revised health literacy-based consent process. J Patient Saf. 2011 Mar;7(1):30-8. doi: 10.1097/PTS.0b013e31820cd632. PMID 21921865
- [Background] Ronco M, Iona L, Fabbro C, Bulfone G, Palese A. Patient education outcomes in surgery: a systematic review from 2004 to 2010. Int J Evid Based Healthc. 2012 Dec;10(4):309-23. doi: 10.1111/j.1744-1609.2012.00286.x. PMID 23173656
- [Background] Gürhan, N., Yaman Sözbir, Ş., & Polat, Ü. (2020). Hemşirelik Alanında Kullanılan Kavram Beceri ve Modeller
- [Background] Kostekli S, Celik S, Keskin E. Evaluation of the effect of endotracheal aspiration at different head heights on oxygenation of the brain by non-invasive method in intensive care patients. J Clin Nurs. 2022 Jun;31(11-12):1709-1720. doi: 10.1111/jocn.16314. Epub 2022 Mar 31. PMID 35362186
- [Background] Cohen FL. Postsurgical pain relief: patients' status and nurses' medication choices. Pain. 1980 Oct;9(2):265-274. doi: 10.1016/0304-3959(80)90013-5. PMID 7454388
- [Derived] Korkmaz S, Seki Z. Determination of the effect of nursing education given before tympanoplasty surgery on the development of postoperative pain and complications. Pain Manag. 2025 Dec 17:1-13. doi: 10.1080/17581869.2025.2604476. Online ahead of print. PMID 41404828